CLINICAL TRIAL: NCT04515810
Title: Planning Advance Care Together (PACT) to Improve Engagement in Advance Care Planning
Brief Title: Mobile Health Application (PACT) to Improve Engagement in Advance Care Planning
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: RG1121852; R37CA246703 (NIH); NCI-2022-00398 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10849 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2020-08-12; First posted 2020-08-17 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Malignant Solid Neoplasm
Keywords: Advance Care Planning; Advance Directives; End-of-Life; Cancer
MeSH Terms: conditions — Death; Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (PACT) (Experimental): Participants use PACT mHealth app.
  Interventions: Other: Internet-Based Intervention; Other: Questionnaire Administration
- Arm II (standard care) (Active Comparator): Participants engage in standard care with no modifications.
  Interventions: Other: Best Practice; Other: Questionnaire Administration

INTERVENTIONS:
Other: Internet-Based Intervention — Use smartphone application
  Arms: Arm I (PACT)
Other: Best Practice — Engage in standard care
  Other Names: standard of care; standard therapy
  Arms: Arm II (standard care)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial tests a new mobile health application (app) called Planning Advance Care Together (PACT) to help people with cancer talk about and plan for advance care planning (the care they would want if they were unable to communicate) with their loved ones and doctors. The development of the PACT mobile app may help future patients incorporate their social network (typically, but not exclusively, family) into the advance care planning process.

DETAILED DESCRIPTION:
OUTLINE: Patients and support persons are randomized to 1 of 2 arms.

ARM I: Participants use PACT mHealth app.

ARM II: Participants engage in standard care with no modifications.

After completion of study intervention, participants are followed up at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* PATIENT: Diagnosis of poor prognosis advanced cancer defined as locally advanced or metastatic cancer and/or disease progression following at least first line systemic therapy.
* PATIENT: Access to a mobile device; the principal investigator (PI) will ensure that those who have access to a mobile device have access to a mobile device with internet access to ensure they can complete study procedures.
* PATIENT: The ability to provide informed consent.
* PATIENT: Identification and enrollment of a loved support person.
* PATIENT: 18 years of age or older.
* SUPPORT PERSON: The person (family member or friend) whom the patient indicates being a support person.
* SUPPORT PERSON: English speaking.
* SUPPORT PERSON: 18 years of age or older and able to provide informed consent.
* PROVIDER: Current clinical practice and/or research with advanced cancer patients.
* PROVIDER: A history of 3+ years working with advanced cancer patients.
* PROVIDER: 18 years of age or older. Providers across disciplines (e.g., social work, oncology) will be enrolled.

Exclusion Criteria:

* PATIENT: Not fluent in English.
* PATIENT: Severely cognitively impaired (as measured by Short Portable Mental Status Questionnaire scores of >= 6) to be delivered by trained study research staff during screening.
* PATIENT: Too ill or weak to complete the interviews (as judged by the interviewer).
* PATIENT: Currently receiving hospice at the time of enrollment.
* PATIENT: Children and young adults under age 18.
* PATIENT: Resides outside of the United States.
* SUPPORT PERSON AND PROVIDERS: Resides outside of the United States.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Accrual rates [Patients] | At 3 months post-randomization
  Will assess the percentage of eligible approached patients who consent to enroll in the study
Feasibility: Accrual rates [Support persons] | At 3 months post-randomization
  Will assess the percentage of eligible approached support persons who consent to enroll in the study
Feasibility: Rates of intervention completion [Patients] | At 3 months post-randomization
  Will assess the percentage of enrolled patients who complete the intervention
Feasibility: Rates of intervention completion [Support persons] | At 3 months post-randomization
  Will assess the percentage of enrolled support persons who complete the intervention
Acceptability of the PACT application: Acceptability E-Scale [Patients] | At 3 months post-randomization
  The Acceptability E-Scale is a 6-item scale, scored on a 5-point Likert scale (e.g., 1=very difficult; 5= very easy), with previously demonstrated good internal consistency (Cronbach's alpha=.76), with higher values indicating higher levels of acceptability.
Acceptability of the PACT application: Acceptability E-Scale [Support persons] | At 3 months post-randomization
  The Acceptability E-Scale is a 6-item scale, scored on a 5-point Likert scale (e.g., 1=very difficult; 5= very easy), with previously demonstrated good internal consistency (Cronbach's alpha=.76), with higher values indicating higher levels of acceptability.
Usability of the PACT application: System Usability Scale (SUS) [Patients] | At 3 months post-randomization
  Usability of the PACT application will be assessed among patients using the System Usability Scale (SUS). The SUS is a 10-item scale, scored on a 5-point Lilkert scale (1=strongly disagree; 5=strongly agree), with higher values indicating higher levels of usability
Usability of the PACT application: System Usability Scale (SUS) [Support persons] | At 3 months post-randomization
  Usability of the PACT application will be assessed among support persons using the System Usability Scale (SUS). The SUS is a 10-item scale, scored on a 5-point Lilkert scale (1=strongly disagree; 5=strongly agree), with higher values indicating higher levels of usability
User satisfaction [Patients] | At 3 months post-randomization
  User satisfaction: Patients will engage in an exit interview that assesses their overall satisfaction with the app on a Likert scale ranging from 1-10 (1=not at all satisfied; 10 = extremely satisfied), with higher values indicating higher levels of satisfaction
User satisfaction [Support persons] | At 3 months post-randomization
  User satisfaction: Support persons will engage in an exit interview that assesses their overall satisfaction with the app on a Likert scale ranging from 1-10 (1=not at all satisfied; 10 = extremely satisfied), with higher values indicating higher levels of satisfaction
User engagement as measured by number of views [Patients] | Baseline to 3 months post-intervention
  User engagement will be assessed through tracking of activity (i.e., number of views) over a 3-month period following randomization.
User engagement as measured by number of views [Support persons] | Baseline to 3 months post-intervention
  User engagement will be assessed through tracking of activity (i.e., number of views) over a 3-month period following randomization.
User engagement as measured by time spent on app [Patients] | Baseline to 3 months post-intervention
  User engagement will be assessed through tracking of activity (i.e., time spent on app) over a 3-month period following randomization.
User engagement as measured by time spent on app [Support persons] | Baseline to 3 months post-intervention
  User engagement will be assessed through tracking of activity (i.e., time spent on app) over a 3-month period following randomization.
Change in level of engagement in advance care planning [Patients] | Baseline to 3 months post-intervention
  Patients will be assessed using the reliable and valid Advance Care Planning Engagement Survey: Action Measures. This scale is composed of four sub scales with a total of 18 items. All items are rated on a yes=1 and no=0. Scores can range from 0 (no action taken) to 18 (all actions taken).
Change in level of engagement in advance care planning [Patients] | Baseline to 6 months post-intervention
  Patients will be assessed using the reliable and valid Advance Care Planning Engagement Survey: Action Measures. This scale is composed of four sub scales with a total of 18 items. All items are rated on a yes=1 and no=0. Scores can range from 0 (no action taken) to 18 (all actions taken).
Change in level of engagement in advance care planning [Support persons] | Baseline to 3 months post-intervention
  Support persons will be assessed using an adapted support person version of the reliable and valid Advance Care Planning Engagement Survey: Action Measures. This scale is composed of four sub scales with a total of 18 items. All items are rated on a yes=1 and no=0. Scores can range from 0 (no action taken) to 18 (all actions taken).
Change in level of engagement in advance care planning [Support persons] | Baseline to 6 months post-intervention
  Support persons will be assessed using an adapted support person version of the reliable and valid Advance Care Planning Engagement Survey: Action Measures. This scale is composed of four sub scales with a total of 18 items. All items are rated on a yes=1 and no=0. Scores can range from 0 (no action taken) to 18 (all actions taken).
Change in documentation of advance care planning conversations [Patients] | Baseline to 3 months post-intervention
  This will be measured using our previously utilized 8-item measure of discussing EoL care, living will, HCP, and DNR orders with family and doctor (all yes/no questions).
Change in documentation of advance care planning conversations [Patients] | Baseline to 6 months post-intervention
  This will be measured using our previously utilized 8-item measure of discussing EoL care, living will, HCP, and DNR orders with family and doctor (all yes/no questions).
Change in documentation of advance care planning conversations [Support persons] | Baseline to 3 months post-intervention
  This will be measured using our previously utilized 8-item measure of discussing EoL care, living will, HCP, and DNR orders with patient and patient's doctor) (all yes/no questions).
Change in documentation of advance care planning conversations [Support persons] | Baseline to 6 months post-intervention
  This will be measured using our previously utilized 8-item measure of discussing EoL care, living will, HCP, and DNR orders with patient and patient's doctor) (all yes/no questions).
Change in completion of advance directives | Baseline to 3 months post-intervention
  This will be assessed by asking patients whether they have completed a Do Not Resuscitate order (DNR), living will, or identified a Health Care Proxy (HCP). All yes/no questions.
Change in completion of advance directives | Baseline to 6 months post-intervention
  This will be assessed by asking patients whether they have completed a Do Not Resuscitate order (DNR), living will, or identified a Health Care Proxy (HCP). All yes/no questions.

SECONDARY OUTCOMES:
Change in treatment preference | Baseline to 3 months
  This will be assessed in patients with an item used previously in our team's NCI-funded cohort studies that asks patients to express a preference for life-extending versus comfort care (two answer choices).
Change in treatment preference | Baseline to 6 months
  This will be assessed in patients with an item used previously in our team's NCI-funded cohort studies that asks patients to express a preference for life-extending versus comfort care (two answer choices).
Change in healthcare utilization (summary score for total number of healthcare services utilized) | Baseline to 3 months
  This measure will assess patients' receipt of life-prolonging care (number of emergency room visits, hospital admissions, length of stay in the hospital, rates of ICU admission) and use of palliative or hospice care (length and duration of palliative and/or hospice care). A total score will be created for healthcare utilization.
Change in healthcare utilization (summary score for total number of healthcare services utilized) | Baseline to 6 months
  This measure will assess patients' receipt of life-prolonging care (number of emergency room visits, hospital admissions, length of stay in the hospital, rates of ICU admission) and use of palliative or hospice care (length and duration of palliative and/or hospice care). A total score will be created for healthcare utilization.
Change in number of subjects receiving goal-concordant care | Baseline to 3 months
  This will be determined by comparing patients' treatment preferences to treatment received. Patients matching on their desired and received care will be designated as having received goal-concordant care.
Change in number of subjects receiving goal-concordant care | Baseline to 6 months
  This will be determined by comparing patients' treatment preferences to treatment received. Patients matching on their desired and received care will be designated as having received goal-concordant care.
Change in perceived social support | Baseline to 3 months
  This will be assessed among patients and support persons using the Multidimensional Scale of Perceived Social Support (MSPSS). The MSPSS is a 12-item valid and reliable measure of social support from family, friends, and significant other, scored on a 5-point Likert scale (1=strongly disagree; 5=strongly agree), with previously reported excellent internal reliability (Cronbach's α = 0.84 to 0.92).
Change in perceived social support | Baseline to 6 months
  This will be assessed among patients and support persons using the Multidimensional Scale of Perceived Social Support (MSPSS). The MSPSS is a 12-item valid and reliable measure of social support from family, friends, and significant other, scored on a 5-point Likert scale (1=strongly disagree; 5=strongly agree), with previously reported excellent internal reliability (Cronbach's α = 0.84 to 0.92).
Change in family functioning | Baseline to 3 months
  This will be assessed among patients and support persons using the Family Relationship Index (FRI), a scale derived from the Family Environment Scale. FRI consists of 12 true/false items consisting of three subscales (cohesiveness, expressiveness, and conflict resolution) with scores ranging from 1 to 4 with higher scores indicating better family functioning. The FRI is well-validated in cancer patients.
Change in family functioning | Baseline to 6 months
  This will be assessed among patients and support persons using the Family Relationship Index (FRI), a scale derived from the Family Environment Scale. FRI consists of 12 true/false items consisting of three subscales (cohesiveness, expressiveness, and conflict resolution) with scores ranging from 1 to 4 with higher scores indicating better family functioning. The FRI is well-validated in cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Megan J Shen, PhD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (4):
- United States (4):
  - Northwell Health, Manhasset, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karnofsky DA. Determining the extent of the cancer and clinical planning for cure. Cancer. 1968 Oct;22(4):730-4. doi: 10.1002/1097-0142(196810)22:43.0.co;2-h. PMID 5212297
- [Background] Tariman JD, Berry DL, Halpenny B, Wolpin S, Schepp K. Validation and testing of the Acceptability E-scale for web-based patient-reported outcomes in cancer care. Appl Nurs Res. 2011 Feb;24(1):53-8. doi: 10.1016/j.apnr.2009.04.003. Epub 2009 Sep 18. PMID 20974066
- [Background] S. Summers and A. Watt,
- [Background] Borsci S, Federici S, Lauriola M. On the dimensionality of the System Usability Scale: a test of alternative measurement models. Cogn Process. 2009 Aug;10(3):193-7. doi: 10.1007/s10339-009-0268-9. Epub 2009 Jun 30. PMID 19565283
- [Background] Sudore RL, Stewart AL, Knight SJ, McMahan RD, Feuz M, Miao Y, Barnes DE. Development and validation of a questionnaire to detect behavior change in multiple advance care planning behaviors. PLoS One. 2013 Sep 5;8(9):e72465. doi: 10.1371/journal.pone.0072465. eCollection 2013. PMID 24039772
- [Background] Mack JW, Weeks JC, Wright AA, Block SD, Prigerson HG. End-of-life discussions, goal attainment, and distress at the end of life: predictors and outcomes of receipt of care consistent with preferences. J Clin Oncol. 2010 Mar 1;28(7):1203-8. doi: 10.1200/JCO.2009.25.4672. Epub 2010 Feb 1. PMID 20124172
- [Background] Zimet GD, Powell SS, Farley GK, Werkman S, Berkoff KA. Psychometric characteristics of the Multidimensional Scale of Perceived Social Support. J Pers Assess. 1990 Winter;55(3-4):610-7. doi: 10.1080/00223891.1990.9674095. PMID 2280326
- [Background] Kissane DW, McKenzie M, McKenzie DP, Forbes A, O'Neill I, Bloch S. Psychosocial morbidity associated with patterns of family functioning in palliative care: baseline data from the Family Focused Grief Therapy controlled trial. Palliat Med. 2003 Sep;17(6):527-37. doi: 10.1191/0269216303pm808oa. PMID 14526887
- [Background] Edwards B, Clarke V. The validity of the family relationships index as a screening tool for psychological risk in families of cancer patients. Psychooncology. 2005 Jul;14(7):546-54. doi: 10.1002/pon.876. PMID 15546124
- [Background] Brinkman-Stoppelenburg A, Rietjens JA, van der Heide A. The effects of advance care planning on end-of-life care: a systematic review. Palliat Med. 2014 Sep;28(8):1000-25. doi: 10.1177/0269216314526272. Epub 2014 Mar 20. PMID 24651708
- [Background] Garrido MM, Balboni TA, Maciejewski PK, Bao Y, Prigerson HG. Quality of Life and Cost of Care at the End of Life: The Role of Advance Directives. J Pain Symptom Manage. 2015 May;49(5):828-35. doi: 10.1016/j.jpainsymman.2014.09.015. Epub 2014 Dec 11. PMID 25498855
- [Background] Detering KM, Hancock AD, Reade MC, Silvester W. The impact of advance care planning on end of life care in elderly patients: randomised controlled trial. BMJ. 2010 Mar 23;340:c1345. doi: 10.1136/bmj.c1345. PMID 20332506
- [Background] Wright AA, Zhang B, Ray A, Mack JW, Trice E, Balboni T, Mitchell SL, Jackson VA, Block SD, Maciejewski PK, Prigerson HG. Associations between end-of-life discussions, patient mental health, medical care near death, and caregiver bereavement adjustment. JAMA. 2008 Oct 8;300(14):1665-73. doi: 10.1001/jama.300.14.1665. PMID 18840840
- [Background] Garrido MM, Harrington ST, Prigerson HG. End-of-life treatment preferences: a key to reducing ethnic/racial disparities in advance care planning? Cancer. 2014 Dec 15;120(24):3981-6. doi: 10.1002/cncr.28970. Epub 2014 Aug 21. PMID 25145489
- [Background] Dow LA, Matsuyama RK, Ramakrishnan V, Kuhn L, Lamont EB, Lyckholm L, Smith TJ. Paradoxes in advance care planning: the complex relationship of oncology patients, their physicians, and advance medical directives. J Clin Oncol. 2010 Jan 10;28(2):299-304. doi: 10.1200/JCO.2009.24.6397. Epub 2009 Nov 23. PMID 19933909
- [Background] Johnson S, Butow P, Kerridge I, Tattersall M. Advance care planning for cancer patients: a systematic review of perceptions and experiences of patients, families, and healthcare providers. Psychooncology. 2016 Apr;25(4):362-86. doi: 10.1002/pon.3926. Epub 2015 Sep 20. PMID 26387480
- [Background] Singer PA, Martin DK, Lavery JV, Thiel EC, Kelner M, Mendelssohn DC. Reconceptualizing advance care planning from the patient's perspective. Arch Intern Med. 1998 Apr 27;158(8):879-84. doi: 10.1001/archinte.158.8.879. PMID 9570174
- [Background] Houben CHM, Spruit MA, Groenen MTJ, Wouters EFM, Janssen DJA. Efficacy of advance care planning: a systematic review and meta-analysis. J Am Med Dir Assoc. 2014 Jul;15(7):477-489. doi: 10.1016/j.jamda.2014.01.008. Epub 2014 Mar 2. PMID 24598477
- [Background] Schobel M, Rieskamp J, Huber R. Social Influences in Sequential Decision Making. PLoS One. 2016 Jan 19;11(1):e0146536. doi: 10.1371/journal.pone.0146536. eCollection 2016. PMID 26784448
- [Background] Pfeiffer E. A short portable mental status questionnaire for the assessment of organic brain deficit in elderly patients. J Am Geriatr Soc. 1975 Oct;23(10):433-41. doi: 10.1111/j.1532-5415.1975.tb00927.x. PMID 1159263
- [Background] Bernard H. Research methods in anthropology: qualitative and quantitative approaches. Lanham, MD: AltaMira; 2005
- [Background] Saunders B, Sim J, Kingstone T, Baker S, Waterfield J, Bartlam B, Burroughs H, Jinks C. Saturation in qualitative research: exploring its conceptualization and operationalization. Qual Quant. 2018;52(4):1893-1907. doi: 10.1007/s11135-017-0574-8. Epub 2017 Sep 14. PMID 29937585
- [Background] Sandelowski M. What's in a name? Qualitative description revisited. Res Nurs Health. 2010 Feb;33(1):77-84. doi: 10.1002/nur.20362. PMID 20014004
- [Background] Sullivan-Bolyai S, Bova C, Harper D. Developing and refining interventions in persons with health disparities: the use of qualitative description. Nurs Outlook. 2005 May-Jun;53(3):127-33. doi: 10.1016/j.outlook.2005.03.005. PMID 15988449
- [Background] Bangor A, Kortum P, Miller J. Determining What Individual SUS Scores Mean: Adding an Adjective Rating Scale. Journal of Usability Studies. 2009;4(3):114-123.
- [Background] Brooke J. SUS: A Retrospective. Journal of Usability Studies. 2013;8(2):29-40.
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] Badr H, Smith CB, Goldstein NE, Gomez JE, Redd WH. Dyadic psychosocial intervention for advanced lung cancer patients and their family caregivers: results of a randomized pilot trial. Cancer. 2015 Jan 1;121(1):150-8. doi: 10.1002/cncr.29009. Epub 2014 Sep 10. PMID 25209975
- [Background] Sobel ME. Asymptotic confidence intervals for indirect effects in structural equation models. Sociological Methodology. 1982;13:290-312.
- [Background] Baron RM, Kenny DA. The moderator-mediator variable distinction in social psychological research: conceptual, strategic, and statistical considerations. J Pers Soc Psychol. 1986 Dec;51(6):1173-82. doi: 10.1037//0022-3514.51.6.1173. PMID 3806354
- [Background] Muller D, Judd CM, Yzerbyt VY. When moderation is mediated and mediation is moderated. J Pers Soc Psychol. 2005 Dec;89(6):852-63. doi: 10.1037/0022-3514.89.6.852. PMID 16393020
- [Background] Preacher KJ, Rucker DD, Hayes AF. Addressing Moderated Mediation Hypotheses: Theory, Methods, and Prescriptions. Multivariate Behav Res. 2007 Jan-Mar;42(1):185-227. doi: 10.1080/00273170701341316. PMID 26821081
- See also: Usability.gov. System Usability Scale (SUS) — https://www.usability.gov/how-to-and-tools/methods/system-usability-scale.html
- See also: Measuring Usability with the System Usability Scale — https://measuringu.com/sus/